CLINICAL TRIAL: NCT02999217
Title: The Impact of Treatment of Anaemia With Intravenous Iron on Haematological Values for Patients After Colorectal Surgery
Brief Title: Intravenous Iron for Correction of Anaemia After Colorectal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaunas University of Medicine (Other)
Collaborators: Orivas, Lithuania (Unknown); Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEC-MF-74
Record Dates: First submitted 2016-10-27; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Anemia, Iron-Deficiency; Intravenous Drug Usage; Colorectal Neoplasms; Colorectal Surgery
Keywords: iron isomaltoside; plasma ferritin; haemoglobin; colorectal cancer
MeSH Terms: conditions — Anemia, Iron-Deficiency; Colorectal Neoplasms | interventions — iron isomaltoside 1000; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): 1 g of intravenous iron isomaltoside given postoperatively for patients with preoperative anaemia (Hb 90-120 g/l and plasma ferritin<100 mkg/l).
  Interventions: Drug: Iron isomaltoside
- Control (Placebo Comparator): The same amount of intravenous saline for patients with preoperative anaemia (Hb 90-120 g/l and plasma ferritin<100 mkg/l).
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Iron isomaltoside — Intravenous injection 1 g given postoperatively in the recovery ward.
  Blood tests including red blood cell count, plasma ferritin, haemoglobin, haematocrit, mean corpuscular volume, mean haemoglobin concentration are made 1 day preoperatively, day 1, day 3 postoperatively, day of discharge and 1 month after discharge.
  Reticulocyte count and reticulocyte haemoglobin concentration tests are made on the day of discharge and 1 month after discharge.
  Count of total consumption of intravenous blood products. Count of total intravenous fluids. Clinical recovery and complications. Duration of hospital stay.
  Other Names: Monofer
  Arms: Treatment
Drug: Saline — Intravenous injection given postoperatively in the recovery ward.
  Blood tests including red blood cell count, plasma ferritin, haemoglobin, haematocrit, mean corpuscular volume, mean haemoglobin concentration are made 1 day preoperatively, day 1, day 3 postoperatively, day of discharge and 1 month after discharge.
  Reticulocyte count and reticulocyte haemoglobin concentration tests are made on the day of discharge and 1 month after discharge.
  Count of total consumption of intravenous blood products. Count of total intravenous fluids. Clinical recovery and complications. Duration of hospital stay.
  Other Names: Sodium chloride
  Arms: Control

SUMMARY:
This 4-week prospective double blind anaemia management study evaluates the effect of high-dose postoperative intravenous iron vs placebo for patients after colorectal cancer surgery. Patients with preoperative levels of haemoglobin 90-120 g/l will be randomly assigned to receive either 1 g of intravenous iron or equal amount of saline postoperatively. Comparison will be based on the levels of haemoglobin, ferritin and other haematological parameters over time and profile of clinical recovery.

The primary end point is that iron isomaltoside given postoperatively is superior to placebo in terms of increase and stability of levels of haemoglobin and other haematological parameters.

DETAILED DESCRIPTION:
The Aim: to assess the effect of treatment of preoperative anaemia with intravenous iron on haematological parameters for patients after elective colorectal surgery.

Primary Hypothesis: postoperative treatment with intravenous iron increases the levels of haemoglobin, ferritin, red cell count and is superior compared to placebo.

Secondary effects: treatment with intravenous iron vs placebo provides reduction of blood transfusions, postoperative complications and hospital stay.

The Objectives:

1. To estimate the rate of preoperative anaemia in patients of elective colorectal surgery.
2. To assess the dynamic changes of total blood count values in colorectal surgery patients treated with postoperative intravenous iron.
3. To compare the changes in total blood count values over time in colorectal surgery patients treated with intravenous iron versus colorectal surgery patients of the control group.

Methods:

The prospective, double-blinded study includes American Society of Anaesthesiology (ASA) I-III patients, aged 18-75 years, admitted for elective colorectal surgery. Preoperatively, patients with levels of haemoglobin 90-120 g/l will be identified and their serum ferritin will be tested. In cases of ferritin<100 mkg/l, patients will be blindly randomized into one of the two groups: treatment group (group T) is given 1000 mg of intravenous iron (iron isomaltoside, Orivas, Pharmacosmos) in the postoperative recovery ward and control group (group C) which is given the same volume of intravenous saline (placebo).

Patients in both groups will be provided with general anaesthesia (fentanyl, propofol, atracurium, inhaled sevoflurane for maintenance) and after tracheal extubation will be transferred to the recovery ward.

Patient blood tests: total blood count, haemoglobin, haematocrit, mean corpuscular volume (MCV), mean corpuscular haemoglobin (MCH), plasma ferritin) will be assessed in both groups 1 day preoperatively, day 1 and 3 postoperatively, the day of discharge and 4 weeks after discharge from the department of surgery. The level of reticulocyte and reticulocyte haemoglobin concentration will be determined on the day of discharge and 4 weeks after discharge.

According to the study protocol, groups will also be compared in terms of clinical recovery, requirements of intravenous fluids and blood transfusion and duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* elective colorectal cancer surgery
* preoperative haemoglobin 90-120 g/l
* preoperative plasma ferritin <100 mkg/l

Exclusion Criteria:

* laparoscopic colorectal surgery
* body mass <50kg
* history of overdosage of iron products
* family history of haemochromatosis, thalassaemia,
* non-iron deficiency anaemia (Vit. B12, folic acid defficiency, haemoglobinopathies)
* under treatment with erythropoietin, intravenous iron or blood transfusion in the last 12 weeks
* allergy to iron carboxymaltose or its supplements
* body temperature > 37.5 °C or under antibiotic use
* chronic liver diseases or/and increased levels of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 3 times over normal upper limit
* patients ill with grave bronchial asthma
* patients with manifestation of allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Changes in haemoglobin level | 4 weeks after surgery
  Haemoglobin level will be tested in both groups at day 1, 3 postoperatively, day of discharge and 4 weeks after surgery

SECONDARY OUTCOMES:
Changes of plasma ferritin | 4 weeks after surgery
  Other haematological variables will be tested in both groups at day 1, 3 postoperatively, day of discharge and 4 weeks after surgery
Changes of red blood cell count | 4 weeks after surgery
  Other haematological variables will be tested in both groups at day 1, 3 postoperatively, day of discharge and 4 weeks after surgery
Changes of mean corpuscular volume | 4 weeks after surgery
  Other haematological variables will be tested in both groups at day 1, 3 postoperatively, day of discharge and 4 weeks after surgery
Changes of mean corpuscular haemoglobin concentration | 4 weeks after surgery
  Other haematological variables will be tested in both groups at day 1, 3 postoperatively, day of discharge and 4 weeks after surgery
Changes of reticulocyte count | 4 weeks after surgery
  It will be tested in both groups at the day of discharge and 4 weeks after surgery
Changes of reticulocyte haemoglobin count | 4 weeks after surgery
  It will be tested in both groups at the day of discharge and 4 weeks after surgery
Rate of blood transfusion | From date of randomization until the day of discharge from the hospital, up to 2 weeks after surgery
  Total amount of blood transfusion units will be counted 2 weeks after surgery in both groups.
Amount of intravenous fluid therapy | From date of randomization until the day of discharge, up to 2 weeks after surgery
  Total amount of intravenous fluids will be counted starting from the date of randomization, separately in the operating room, recovery area and each day postoperatively until 2 weeks after surgery in both groups.
Number of participants with perioperative complications | 4 weeks after surgery
  Total number of postoperative complications will be counted in both groups.
Duration of hospital stay | From the date of randomization until the day of discharge, up to 2 weeks after surgery
  It will be counted in both groups 2 weeks after surgery in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andrius Macas, MDPhDProf, Study Chair — Head of the Department of Anaesthesiology, Medical academy, Lithuanian University of Health Sciences
Locations (1):
- Department of Anaesthesiology, Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available within 6 months of study completion.

REFERENCES:
- [Background] Shander A, Knight K, Thurer R, Adamson J, Spence R. Prevalence and outcomes of anemia in surgery: a systematic review of the literature. Am J Med. 2004 Apr 5;116 Suppl 7A:58S-69S. doi: 10.1016/j.amjmed.2003.12.013. PMID 15050887
- [Background] Edna TH, Karlsen V, Jullumstro E, Lydersen S. Prevalence of anaemia at diagnosis of colorectal cancer: assessment of associated risk factors. Hepatogastroenterology. 2012 May;59(115):713-6. doi: 10.5754/hge11479. PMID 22469713
- [Background] Ward DG, Roberts K, Brookes MJ, Joy H, Martin A, Ismail T, Spychal R, Iqbal T, Tselepis C. Increased hepcidin expression in colorectal carcinogenesis. World J Gastroenterol. 2008 Mar 7;14(9):1339-45. doi: 10.3748/wjg.14.1339. PMID 18322945
- [Background] Ganz T. Hepcidin and iron regulation, 10 years later. Blood. 2011 Apr 28;117(17):4425-33. doi: 10.1182/blood-2011-01-258467. Epub 2011 Feb 23. PMID 21346250
- [Background] Leichtle SW, Mouawad NJ, Lampman R, Singal B, Cleary RK. Does preoperative anemia adversely affect colon and rectal surgery outcomes? J Am Coll Surg. 2011 Feb;212(2):187-94. doi: 10.1016/j.jamcollsurg.2010.09.013. PMID 21276532
- [Background] Cladellas M, Bruguera J, Comin J, Vila J, de Jaime E, Marti J, Gomez M. Is pre-operative anaemia a risk marker for in-hospital mortality and morbidity after valve replacement? Eur Heart J. 2006 May;27(9):1093-9. doi: 10.1093/eurheartj/ehi830. Epub 2006 Mar 14. PMID 16537556
- [Background] Hogan M, Klein AA, Richards T. The impact of anaemia and intravenous iron replacement therapy on outcomes in cardiac surgery. Eur J Cardiothorac Surg. 2015 Feb;47(2):218-26. doi: 10.1093/ejcts/ezu200. Epub 2014 May 13. PMID 24824650
- [Background] Elhenawy AM, Meyer SR, Bagshaw SM, MacArthur RG, Carroll LJ. Role of preoperative intravenous iron therapy to correct anemia before major surgery: study protocol for systematic review and meta-analysis. Syst Rev. 2015 Mar 15;4:29. doi: 10.1186/s13643-015-0016-4. PMID 25874460